CLINICAL TRIAL: NCT07373197
Title: Lateral Rectus Muscle Strangulation: A New Weakening Technique in Cases of Exotropia
Brief Title: Lateral Rectus Muscle Strangulation in Cases of Exotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Mounir, Assistant Professor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-09-12PD
Record Dates: First submitted 2025-09-25; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Strabismus, Divergent
Keywords: Exotropia; Lateral rectus muscle
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lateral rectus muscle strangulation (Experimental): lateral rectus muscle strangulation as a weakening technique in cases of exotropia.
  Interventions: Procedure: Muscle strangulation

INTERVENTIONS:
Procedure: Muscle strangulation — lateral rectus muscle strangulation as a weakening technique in cases of exotropia.

SUMMARY:
The goal of our study to evaluate effect of lateral rectus muscle strangulation as a novel effective weakening technique in cases of exotropia.

It is a case-series intervensional study with a total 12 participant who are diagnosed as exophoria or intermittent exotropia who are older than 4 years old.

All patients will be assessed regarding their angle of deviation and then undergo lateral rectus muscle strangulation under general anesthesia and then will be followed- up at 1st day, 1st week, 1st month and 6th months.

DETAILED DESCRIPTION:
Under general anesthesia and after sterilization and draping of the eyes, an eye speculum is inserted. The muscle is exposed and hooked through either a fornix-based or limbal-based incision. Careful dissection is carried out to delineate the muscle edge, a previously measured blook of the lateral rectus muscle is sutured (strangulated) with proline 10/0 as in (fig-1). Patients will be followed-up next day after surgery then after 1 month and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* intermittent exotropia

Exclusion Criteria:

* previous squint surgery

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Correction of strabismus | 12 months
  the correction was done by lateral rectus muscle strangulation

SECONDARY OUTCOMES:
orthophoria | 12 months
  to make both eyes aligned together, and to maintain orthophoria

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
we havenot decided until now to share IPD with other researchers

REFERENCES:
- [Background] Rageh MA, Awadein A, Arfeen SA. Extraocular muscle fenestration: a novel weakening procedure. Can J Ophthalmol. 2020 Oct;55(5):455-457. doi: 10.1016/j.jcjo.2020.05.018. Epub 2020 Aug 26. No abstract available. PMID 32860744
- [Background] Taher SG, Rageh MA, Hashem O. Extra Ocular Muscle Fenestration as a Weakening Maneuver for Surgical Management of Strabismus: A Randomized Pilot Clinical Trial. Clin Ophthalmol. 2022 Jan 8;16:63-70. doi: 10.2147/OPTH.S347092. eCollection 2022. PMID 35035214
- [Background] Koc F, Ozal H, Yasar H, Firat E. Resolution in partially accomodative esotropia during occlusion treatment for amblyopia. Eye (Lond). 2006 Mar;20(3):325-8. doi: 10.1038/sj.eye.6701874. PMID 15933753
- See also: Related Info — https://www.healthline.com/health/exophoria

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07373197/Prot_SAP_000.pdf